CLINICAL TRIAL: NCT05004129
Title: An Open-Label Study to Evaluate the Long-Term Safety and Efficacy of Tideglusib for the Treatment of Congenital or Childhood Onset DM1 (REACH CDM X)
Brief Title: Safety and Efficacy of Tideglusib in Congenital or Childhood Onset Myotonic Dystrophy
Acronym: REACH CDM X
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AMO Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMO-02-MD-2-004
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Congenital Myotonic Dystrophy
Keywords: Tideglusib; AMO-02-MD-2-004; Congenital Myotonic Dystrophy; Myotonic Dystrophy; Dystrophia Myotonica; Myotonia Atrophica; Myotonia Dystrophica; Myotonic Dystrophy, Congenital; Steinert Disease; Steinert Myotonic Dystrophy; Steinert's Disease
MeSH Terms: conditions — Myotonic Dystrophy | interventions — tideglusib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tideglusib (Experimental): Weight adjusted or weight banded tideglusib, orally, once daily
  Interventions: Drug: Tideglusib

INTERVENTIONS:
Drug: Tideglusib — Tideglusib dosing will be weight-adjusted at 400 mg, 600 mg, or 1000 mg dose levels, or weight banded fixed doses of 400 mg, 600 mg, 800 mg or 1000 mg, with each subject starting at a weight-adjusted 400 mg dose level for 2 weeks, then up titrating to a weight-adjusted 600 mg dose level for the next 2 weeks.

SUMMARY:
This is an open-label phase 2/3 study for individuals with Congenital Myotonic Dystrophy (Congenital DM1) who participated in the preceding AMO-02-MD-2-003 study or individuals with either Congenital or Childhood Onset DM1 who are treatment naïve.

DETAILED DESCRIPTION:
This is an open-label study of either a weight-adjusted 1000 mg fixed dose or a weight banded fixed dose of tideglusib across a 52-week treatment period with an open-ended optional extended access period. The subjects are children and adolescents with Congenital DM1 who participated in the antecedent AMO-02-MD-2-003 study or individuals with either Congenital or Childhood onset DM1 who are treatment naïve.

ELIGIBILITY:
Inclusion Criteria:

Subjects who do not enter this study directly from completing the AMO-02-MD-2-003 study (i.e. subjects who did not complete AMO-02-MD-2-003, subjects who completed AMO-02-MD-2-003 but did not directly rollover or subjects who are re-entering AMO-02-MD-2-004), will not be considered eligible for the study without meeting all of the criteria below:

1. Subjects under study must be individuals with a diagnosis of Congenital or Childhood Onset DM1.
2. Diagnosis must be genetically confirmed
3. Subjects must be male or female aged ≥6 years to ≤45 years at Screening
4. Subjects must have a Clinical Global Impression - Severity (CGI-S) score of 3 or greater at Screening (V-1)
5. Written, voluntary informed consent must be obtained before any study related procedures are conducted. Where a parent or legally authorized representative (LAR) provides consent, there must also be assent from the subject (as required by local regulations)
6. Subject's caregiver must be willing and able to support participation for duration of study
7. Subject must be willing and able to comply with the required food intake restrictions as outlined per protocol

Subjects entering directly from completing the antecedent AMO-02-MD-2-003 study will not be considered eligible for the study without meeting all of the criteria below:

1. Subjects who have completed the antecedent AMO-02-MD-2-003 study through V11
2. Written, voluntary informed consent must be obtained before any study related procedures are conducted. Where a parent or LAR provides consent, there must also be assent from the subject (as required by local regulations)
3. Subject's caregiver must be willing and able to support participation for duration of study
4. Subject must be willing and able to comply with the required food intake restrictions as outlined per protocol

Key Exclusion Criteria:

1. Body mass index (BMI) less than 13.5 kg/m² or greater than 40 kg/m²
2. New or change in medications/therapies within 4 weeks prior to Eligibility/Baseline Visit
3. Use within 4 weeks prior to Eligibility/Baseline Visit of strong CYP3A4 inhibitors (eg.clarithromycin, telithromycin, ketoconazole, itraconazole, posaconazole, nefazodone, idinavir and ritonavir)
4. Concurrent use of drugs metabolized by CYP3A4 with a narrow therapeutic window (e.g. warfarin and digitoxin)
5. Current enrollment in a clinical trial of an investigational drug or enrollment in a clinical trial of an investigational drug in the last 6 months other than the AMO-02- MD-2-003 study
6. Existing or historical medical conditions or complications (eg. neurological, cardiovascular, renal, hepatic, gastrointestinal, endocrine or respiratory disease) that may impact the interpretability of the study results
7. Hypersensitivity to tideglusib or any components of its formulation including allergy to strawberry

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety (Adverse Events) | 52 Weeks
  The incidence of AEs, including SAEs, and abnormal findings in objective assessments (e.g. laboratory values, ECGs and vital signs) from Screening to Enrolment (where applicable), from Enrolment to End of Treatment (52 Weeks), and End of Treatment to the End of Follow-up period.
Safety (Adverse Events) - With Optional Expanded Access | Week 60 and every 8 weeks thereafter up until discontinuation or study closure, assessed up to Week 132
  The incidence of AEs, including SAEs, and abnormal findings in objective assessments (e.g. laboratory values, ECGs and vital signs) from End of Treatment to End of Optional Extended Access, and End of Optional Extended Access to the End of Follow-up period.
Clinician-Completed Congenital DM1 Rating Scale (CDM1-RS) | 52 Weeks
  The Clinician-completed Congenital DM1 Rating Scale is an 11-item rating scale completed by the clinician to score the symptom severity of domains that are clinically relevant in Congenital DM1.

SECONDARY OUTCOMES:
Clinician-Completed Congenital DM1 Rating Scale (CDM1-RS) - With Optional Expanded Access | Week 68 and every 16 weeks thereafter up until discontinuation or study closure, assessed up to Week 132
  The Clinician-completed Congenital DM1 Rating Scale is an 11-item rating scale completed by the clinician to score the symptom severity of domains that are clinically relevant in Congenital DM1.
Clinical Global Impressions Improvement Scale (CGI-I) | 54 Weeks
  The CGI-I requires the clinician to rate how much the subject's illness has changed (improved, worsened or stayed the same) relative to a baseline state.
Clinical Global Impressions Improvement Scale (CGI-I) - With Optional Expanded Access | Week 68 and every 16 weeks thereafter up until discontinuation or study closure, assessed up to Week 132
  The CGI-I requires the clinician to rate how much the subject's illness has changed (improved, worsened or stayed the same) relative to a baseline state.
Top 3 Caregiver Concerns Visual Analogue Scale (VAS) score | 54 weeks
  The Top 3 concerns VAS allows caregivers to identify their main three causes of concern, related to the subject's myotonic dystrophy, rather than these being pre-specified within a scale and then rating how these concerns have changed at specific time-points during the study.
Top 3 Caregiver Concerns Visual Analogue Scale (VAS) score - With Optional Expanded Access | Week 68 and every 16 weeks thereafter up until discontinuation or study closure, assessed up to Week 132
  The Top 3 concerns VAS allows caregivers to identify their main three causes of concern, related to the subject's myotonic dystrophy, rather than these being pre-specified within a scale and then rating how these concerns have changed at specific time-points during the study.
Caregiver Completed Congenital DM1 Rating Scale (CC-CDM1-RS) | 52 weeks
  CC-CDM1-RS provides a caregiver assessment of the subject on symptoms that may occur in individuals with CDM1. There are a total of 11 symptoms that the caregiver is asked to rate from 0 to 4 based on overall severity.
Caregiver Completed Congenital DM1 Rating Scale (CC-CDM1-RS) - With Optional Expanded Access | Week 68 and every 16 weeks thereafter up until discontinuation or study closure, assessed up to Week 132
  CC-CDM1-RS provides a caregiver assessment of the subject on symptoms that may occur in individuals with CDM1. There are a total of 11 symptoms that the caregiver is asked to rate from 0 to 4 based on overall severity.
Clinical Global Impressions Severity Scale (CGI-S) | 54 weeks
  The CGI-S is a 7-point Likert type scale that requires the clinician to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis.
Clinical Global Impressions Severity Scale (CGI-S) - With Optional Expanded Access | Week 68 and every 16 weeks thereafter up until discontinuation or study closure, assessed up to Week 132
  The CGI-S is a 7-point Likert type scale that requires the clinician to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis.
Autism Behavior Inventory- Clinician (ABI-C) | 52 Weeks
  ABI-C is a 14 item rating scale requires the clinician to assess the core features of Autism Spectrum Disorder as well as common associated behaviors.
Socialization, Communication, Daily Living, and Adaptive Behavior Composite standard scores of the Vineland Adaptive Behavior Scale - Survey Interview | 52 Weeks
  The Vineland Adaptive Behavior Scales require the clinician to measure personal and social skills needed for everyday living. It provides a targeted assessment of adaptive behavior via a semi-structured parent or caregiver interview.
10-meter walk-run test | 52 Weeks
  The 10-meter walk/run test is a performance measure used to assess walking speed in meters per second over a short distance. It can be used as an assessment of functional mobility.
Plasma Troponin T levels | 52 Weeks
  Troponin T can be used as a biomarker for cardiac dysfunction but can also be elevated in DM1 patients without evident cardiac dysfunction.
Plasma Troponin T levels - With Optional Expanded Access | Week 68 and every 16 weeks thereafter up until discontinuation or study closure, assessed up to Week 132
  Troponin T can be used as a biomarker for cardiac dysfunction but can also be elevated in DM1 patients without evident cardiac dysfunction.
Blood Leukocytes CTG Repeats | Baseline and Week 52
  A genomic blood sample will be taken from all subjects to confirm the average number of repeats at sampling and estimate the number of leukocyte CTG repeats inherited for an individual subject.
Blood Leukocytes CTG Repeats - With Optional Expanded Access | Week 52 or later
  A genomic blood sample will be taken from all subjects to confirm the average number of repeats at sampling and estimate the number of leukocyte CTG repeats inherited for an individual subject. For subjects that have already passed Week 52 at implementation of this endpoint, a single genomic blood sample will taken at the next in-clinic OEA visit.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Gray-Stephens, BM BCh, MA (Oxon), MFPM, Study Director — AMO Pharma
Locations (14):
- United States (10):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Palo Alto, California
  - Lurie's Children's Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Rochester - Medical Center, Rochester, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University-Department of Neurology - Muscular Dystrophy Translational Research Program, Richmond, Virginia
- The Bright Alliance, Randwick, New South Wales, Australia
- Canada (2):
  - Children's Hospital London Health Sciences Centre (LHSC), London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
- New Zealand Clinical Research (NZCR), Auckland, New Zealand